CLINICAL TRIAL: NCT03995459
Title: Deportalization, Venous Deprivation, Venous Congestion: Impact on Liver Volume and Function
Brief Title: Deportalization, Venous Deprivation, Venous Congestion
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0250
Record Dates: First submitted 2019-06-03; First posted 2019-06-24 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Malignant Liver Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with multiple primary or secondary liver tumors have a low survival rate unless they can benefit from curative extended hepatic resections with R0 or R1 marge resection. Post-operative acute liver failure may occur after such surgery when the remnant liver is insufficient, leading to high morbimortality.

The future remnant liver (FRL) preoperative evaluation is then the key consideration before performing extended liver resection. The FRL volume measurement on computed tomography (CT) imaging is the most widespread method of FRL evaluation. Threshold values of acceptable FRL volume depend on the underlying liver function, it ranges from 20-30% in healthy liver to 40% in cirrhotic liver. However, it recently appeared that the FRL function would be more valuable in predicting post-operative liver failure. 99mTc-mebrofenin hepatobiliary scintigraphy (HBS) combined with SPECT/CT enables reliable FRL function measurement with a threshold value calculated at 2.69%/min/m2, to predict post-hepatectomy liver failure.

When the FRL evaluation does not reach the acceptable threshold values to avoid liver failure, portal vein embolization (PVE), consisting of portal branches occlusion of the future removed liver, can be performed. It is now the standard of care to induce FRL regeneration before surgery. Right PVE induces right hemiliver (S5-8) deportalization (portal input deprivation with hepatic venous drainage preservation) leading to left hemiliver (S2-4) regeneration.

To optimize PVE results, recent effective techniques have been developed such as the simultaneous embolization of the right portal branch and the right hepatic vein (HV), and the right accessory HV if so, which is called liver venous deprivation technique. Additional simultaneous embolization of the middle HV defined the extended liver venous deprivation (ELVD) technique. ELVD induces right liver (S5-8) venous deprivation (deprivation of both portal input and venous drainage) and leads to rapid increase in FRL function. After ELVD, segment IV (S4) portal input from left portal branch is preserved while its venous drainage through the middle HV is disrupted, resulting in venous congestion.

The aim of this study is to analyze the volumetric and functional evolutions after embolization procedures in deportalized liver (S5-8 after PVE), vein-deprived liver (S5-8 after ELVD) and congestive liver (S4 after ELVD).

ELIGIBILITY:
Inclusion criteria:

* Age > or = 18 years
* primary or secondary liver tumor(s)
* major hepatectomy approved by multidisciplinary tumor meeting
* small FRL (baseline FLR <2.69%/min/m2)

Exclusion criteria:

* liver fibrosis / cirrhosis
* biliary obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the investigator's institution for major hepatectomy in a context of small FLR. Small FRL was defined as baseline FLR function (clearance rate of 99mTc-mebrofenin) <2.69%/min/m2
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline liver volume | day 7, day 14 and day 21
  1. Change from baseline liver volume (expressed in mL, assessed by manual regional volumetric measurements on CT) in the deportalized liver, the vein deprived liver and the congestive liver at day 7, day 14 and day 21.
Evolution from baseline of liver volume and liver function values | 1 day
  Evolution from baseline of liver volume and liver function values in the deportalized liver, the vein deprived liver and the congestive liver respectively : liver function (%/min/m2): assessed by regional measurements on 99mTC-mebrofenin hepatobiliary scintigraphy

SECONDARY OUTCOMES:
Evolution from baseline of liver volume and liver function values | day 7, day 14 and day 21
  Evolution from baseline of liver volume and liver function values in the non embolized liver : liver volume (mL): assessed by manual regional volumetric measurements on CT at baseline, day 7, day 14 and day 21
Evolution from baseline of liver volume and liver function values | 1 day
  Evolution from baseline of liver volume and liver function values in the non embolized liver : liver function (%/min/m2): assessed by regional measurements on 99mTC-mebrofenin hepatobiliary scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC